CLINICAL TRIAL: NCT05107674
Title: A Phase 1a, Dose Escalation, Safety and Tolerability Study of NX-1607, a Casitas B-lineage Lymphoma Proto-oncogene (CBL-B) Inhibitor, in Adults With Advanced Malignancies, With Phase 1b Expansion in Select Tumor Types
Brief Title: A Study of NX-1607 in Adults With Advanced Malignancies
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Nurix Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NX-1607-101
Record Dates: First submitted 2021-09-22; First posted 2021-11-04 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Ovarian Cancer, Epithelial; Gastric Cancer; GastroEsophageal Junction (GEJ) Cancer; Head and Neck Squamous Cell Carcinoma; Metastatic or Unresectable Melanoma; Non-small Cell Lung Cancer (NSCLC); Metastatic Castration-resistant Prostate Cancer (mCRPC); Malignant Pleural Mesothelioma (MPM); Triple Negative Breast Cancer (TNBC); Metastatic Urothelial Carcinoma; Cervical Cancer; Diffuse Large B Cell Lymphoma (DLBCL); Richter Transformation; Microsatellite Stable Colorectal Carcinoma
Keywords: Ubiquitin Ligase Inhibitor; Advanced Malignancies; T-cell Activation
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Stomach Neoplasms; Neoplasms; Squamous Cell Carcinoma of Head and Neck; Neoplasm Metastasis; Carcinoma, Non-Small-Cell Lung; Mesothelioma, Malignant; Triple Negative Breast Neoplasms; Carcinoma, Transitional Cell; Uterine Cervical Neoplasms; Lymphoma, Large B-Cell, Diffuse | interventions — Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (12):
- Phase 1a Dose Escalation of NX-1607 (monotherapy) (Experimental): Multiple dose levels and dosing regimen of NX-1607 to be evaluated; determination of MTD/Phase 1b recommended dose.
  Interventions: Drug: NX-1607
- Phase 1a Food Effect (Experimental): Impact of food on NX-1607 bioavailability and tolerability to be evaluated
  Interventions: Drug: NX-1607
- Phase 1b Dose Expansion in platinum-resistant EOC (Experimental): Patients with platinum-resistant EOC, including primary peritoneal and fallopian tube carcinoma
  Interventions: Drug: NX-1607
- Phase 1b Dose Expansion in advanced gastric/GEJ cancer (Experimental): Patients with recurrent, locally advanced, or metastatic gastric or GEJ adenocarcinoma
  Interventions: Drug: NX-1607
- Phase 1b Dose Expansion in HNSCC (Experimental): Patients with recurrent, locally advanced, or metastatic HNSCC
  Interventions: Drug: NX-1607
- Phase 1b Dose Expansion in recurrent melanoma (Experimental): Patients with recurrent and either metastatic or unresectable Melanoma
  Interventions: Drug: NX-1607
- Phase 1b Dose Expansion in advanced NSCLC (Experimental): Patients with Stage IV NSCLC
  Interventions: Drug: NX-1607
- Phase 1b Dose Expansion in mCRPC (Experimental): Patients with mCRPC who received a minimum of 2 prior lines of therapy in the advanced setting including androgen receptor-directed therapy and a taxane-based chemotherapy and has PSA or radiographic progression
  Interventions: Drug: NX-1607
- Phase 1b Dose Expansion in mixed solid tumor cohort (Experimental): Cohort of mixed solid tumor indications consisting of patients with MPM, TNBC, locally advanced or metastatic urothelial cancer, cervical cancer, or DLBCL/DLBCL-RT
  Interventions: Drug: NX-1607
- Phase 1a Dose Escalation of NX-1607 in combination with Paclitaxel (Experimental): Indications may include but are not limited to, platinum resistant EOC, gastric/GEJ cancer. HSNCC, NSCLC, TNBC, locally advanced or metastatic urothelial cancer and cervical cancer.
  Interventions: Drug: NX-1607; Drug: Paclitaxel
- Phase 1b Dose Expansion of NX-1607 in combination with Paclitaxel (Experimental): Indications may include but are not limited to, platinum resistant EOC, gastric/GEJ cancer, HSNCC, NSCLC, TNBC, and locally advanced or metastatic urothelial cancer and cervical cancer
  Interventions: Drug: NX-1607; Drug: Paclitaxel
- Phase 1b Dose Expansion in MSS CRC (Experimental): Patients with histologically confirmed MSS CRC, known KRAS WT, and must have been previously treated with > = 2 lines of systemic therapy including a fluoropyrimidine, irinotecan, and/or oxaliplatin (and EGFR inhibitor if known Ras wild type)
  Interventions: Drug: NX-1607

INTERVENTIONS:
Drug: NX-1607 — Oral NX-1607
  Other Names: Cbl-b Inhibitor
Drug: Paclitaxel — Paclitaxel IV
  Arms: Phase 1a Dose Escalation of NX-1607 in combination with Paclitaxel; Phase 1b Dose Expansion of NX-1607 in combination with Paclitaxel

SUMMARY:
This is a first-in-human Phase 1a/1b multicenter, open-label oncology study designed to evaluate the safety and anti-cancer activity of NX-1607 in patients with advanced malignancies.

DETAILED DESCRIPTION:
Phase 1a will consist of 2 study arms: Monotherapy and Paclitaxel combo. Phase 1a dose escalation will evaluate the safety and tolerability of NX-1607 in adult patients with advanced solid tumors for which standard therapy with proven clinical benefit does not exist, is no longer effective, or is not appropriate. Indications for monotherapy include platinum resistant epithelial ovarian cancer (EOC), gastric/gastroesophageal junction (GEJ) cancer, squamous cell carcinoma of the head and neck (HNSCC), recurrent and either metastatic or unresectable melanoma, non-small cell lung cancer (NSCLC), metastatic castration-resistant prostate cancer (mCRPC), malignant pleural mesothelioma (MPM), triple-negative breast cancer (TNBC), locally advanced or metastatic urothelial cancer, cervical cancer, and microsatellite stable colorectal cancer (MSS CRC), and diffuse large cell B-cell lymphoma (DLBCL) including patients with Richter transformation (DLBCL-RT). Indications for paclitaxel combo may include, but are not limited to, platinum-resistant EOC, gastric/GEJ cancer, HNSCC, NSCLC, TNBC, locally advanced or metastatic urothelial cancer, and cervical cancer at the Sponsor's discretion.

Phase 1b will investigate the efficacy of NX-1607 as monotherapy or in combination with paclitaxel at the dose(s) selected in Phase 1a in select advanced malignancies for which standard therapy, including immunotherapy, with proven clinical benefit does not exist, is no longer effective, or is not appropriate. Indications include platinum-resistant EOC, including primary peritoneal and fallopian tube carcinoma, advanced gastric/GEJ cancer, HNSCC, recurrent and either metastatic or unresectable melanoma, advanced NSCLC, mCRPC, MSS CRC, mixed solid tumor cohort indications consisting of patients with MPM, TNBC, locally advanced or metastatic urothelial cancer, cervical cancer, and DLBCL including patients with DLBCL-RT. In Arm 1 (NX-1607 monotherapy), more than 1 dose level of NX-1607 may be tested in individual indications, each of which will constitute a separate cohort in Phase 1b.

ELIGIBILITY:
Key Inclusion Criteria:

* Age ≥ 18 years.
* Measurable disease per disease-specific response criteria.
* Patients must have disease that is metastatic or unresectable and have received standard treatment options, are not candidates for standard treatment options, or will otherwise be prevented from receiving any standard treatment options.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Minimum of 3 weeks or 5 half-lives (whichever is shorter) since last dose of systemic cancer therapy (unless otherwise specified) or minimum of 2 weeks since last radiotherapy, or minimum of 6 weeks since last systemic therapy with nitrosoureas, antibody-drug conjugate, or radio immuno-conjugate therapy.
* Adequate organ and bone marrow function, in the absence of growth factors (with limited exception for DLBCL), as defined by laboratory parameters.
* Patients of child-bearing potential must use adequate contraceptive measures to avoid pregnancy for the duration of the study as defined in the protocol.
* Patient must be willing and able to adhere to the prohibitions and restrictions specified in the protocol.
* Each patient must sign an informed consent form (ICF).
* Histological or cytological diagnosis of platinum-resistant EOC, including primary peritoneal and fallopian tube carcinoma; gastric/GEJ cancer; HNSCC; recurrent and either metastatic or unresectable melanoma; NSCLC; mCRPC; MPM; TNBC; locally advanced or metastatic urothelial cancer; cervical cancer; MSS CRC; or DLBCL (including DLBCL-RT)
* Accessible tumor (for all cohorts) or lymph node (DLBCL only) for biopsy (Phase 1b only).

Key Exclusion Criteria:

* Active untreated brain metastases.
* Patient has any of the following:
* Uncontrolled intercurrent illness including, but not limited to, poorly controlled hypertension or diabetes, or ongoing active infection requiring systemic therapy.
* Patients with primary refractory EOC defined as patients who do not respond to their first platinum-containing regimen or who relapse less than 6 months after completion of that first platinum-containing regimen
* Psychiatric illness that would limit compliance with study requirements.
* Treatment with any of the following prior to the first dose of NX-1607: CPI (anti-PD-1, PD-L1, cytotoxic T-lymphocyte-associated protein 4, etc) within 3 weeks; autologous or allogeneic stem cell transplant within 100 days; prior systemic cancer therapy within 3 weeks or 5 half-lives (whichever is shorter) (unless otherwise specified) (including hormonal therapy except for hormonal prophylaxis for a prior malignancy); prior radiotherapy within 2 weeks; prior systemic therapy with nitrosoureas, antibody-drug conjugate, or radio-immuno-conjugate therapy within 6 weeks; use of strong or moderate CYP3A4 inducers or inhibitors within 14 days or 7 days, respectively, or 5 half-lives (whichever is longer)
* History of CAR-T therapy within 30 days prior to the first dose of NX-1607.
* Toxicities from previous anti-cancer therapies that have not resolved to baseline levels or to Grade 1 or less except for Grade 2 alopecia and Grade 2 peripheral neuropathy or patients receiving endocrine replacement therapy
* Patients who experienced Grade 3 or higher irAEs with prior immunotherapy.
* History of uveitis, or an active autoimmune disease that has required systemic treatment in the past 2 years (i.e., with use of disease modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment and is allowed.
* Unable to swallow capsules or has malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel or ulcerative colitis, symptomatic inflammatory bowel disease, or partial or complete bowel obstruction likely to interfere with the delivery, absorption, or metabolism of NX-1607.
* Known allergies, hypersensitivity, or intolerance to components of NX-1607.
* Pregnant, breastfeeding, or planning to become pregnant while enrolled in this study or within 6 months after the last dose of NX-1607.
* Patient is a man who plans to father a child while enrolled in this study or within 3 months after the last dose of NX-1607 and, as applicable, within 6 months after the last dose of paclitaxel.
* Patient has had major surgery (e.g., requiring general anesthesia) within 4 weeks before the planned first dose of NX-1607, or will not have fully recovered from surgery, or has surgery planned during the time the patient is expected to participate in the study or within 4 weeks after the last dose of NX-1607. Note: Patients with minor planned surgical procedures to be conducted under local anesthesia may participate.
* Vaccinated with a live vaccine within 28 days (with the exception of the annual inactivated influenza vaccine) or COVID-19 vaccination within 14 days prior to the first dose of NX-1607.
* Active known second malignancy with the exception of any of the following:

  * Adequately treated basal cell carcinoma, squamous cell carcinoma of the skin, or in situ cervical cancer.
  * Adequately treated Stage I cancer from which the patient is currently in remission and has been in remission for ≥ 2 years.
  * Low-risk prostate cancer with Gleason score < 7 and PSA < 10 ng/mL.
  * Any other cancer from which the patient has been disease-free for ≥ 2 years.
* Infection with human immunodeficiency virus (HIV)-1 or HIV-2. Exception: Patients with well controlled HIV (e.g., CD4 > 350/mm3 and undetectable viral load) are eligible.
* Current active hepatitis, including hepatitis A (hepatitis A virus immunoglobulin M [IgM] positive), hepatitis B (hepatitis B virus [HBV] surface antigen positive), or hepatitis C (hepatitis C virus [HCV] antibody positive, confirmed by HCV RNA). Patients with HCV with undetectable virus after treatment are eligible. Patients with prior exposure to HBV may be entered if quantitative PCR is negative.
* Use of systemic corticosteroids (> 20 mg prednisone or equivalent) within 15 days (except for prophylaxis for radio diagnostic contrast reactions and/or prophylaxis for patients receiving paclitaxel), or other immunosuppressive drugs within 30 days, prior to the first dose of NX-1607.
* Use of biotin (i.e., Vitamin B7) or supplements containing biotin higher than the daily adequate intake of 30 µg [NIH 2020] (Note: Patients who switch from a high dose to a dose of 30 µg/day or less at least 1 day prior to Screening assessments are eligible for study entry).
* Receipt of an IP or has been treated with an investigational device within 3 weeks or 5 half-lives (whichever is shorter) prior to the first dose of NX-1607.
* Any of the following within 6 months prior to the first dose of NX-1607 or ongoing:

  * Myocardial infarction
  * Unstable angina
  * Unstable symptomatic ischemic heart disease
  * New York Heart Association Class III or IV heart failure
  * Thromboembolic events (e.g., deep vein thrombosis, pulmonary embolism, or symptomatic cerebrovascular events)
  * Any other significant cardiac condition (e.g., pericardial effusion, restrictive cardiomyopathy, severe untreated valvular stenosis, or severe congenital heart disease)
  * Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the participant's participation for the full duration of the study, or is not in the best interest of the participant to participate, in the opinion of the treating Investigator in consultation with the Medical Monitor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 345 (Estimated)
Dates: Start 2021-09-29 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2028-02-28 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs), including Grade ≥ 3 TEAEs, treatment-emergent serious adverse events (SAEs), TEAEs leading to study drug discontinuation, and deaths due to TEAEs | 16 months
  Phase 1a
Incidence of immune-related AEs (irAEs), all deaths, and dose-limiting toxicities (DLTs) | Up to 2 Years
  Phase 1a
Objective Response Rate (ORR) per disease-specific response criteria as assessed by the Investigator | Up to 3 Years
  Phase 1b

SECONDARY OUTCOMES:
PK parameters of NX-1607: area under the curve (AUC) | Up to 3 Years
  Phase 1a/1b - Sampling following the first dose, pre and post-dose at selected cycles, and at the end of treatment
PK parameters of NX-1607: apparent clearance (CL/F) | Up to 3 Years
  Phase 1a/1b - Sampling following the first dose, pre and post-dose at selected cycles, and at the end of treatment
PK parameters of NX-1607: maximum plasma concentration (Cmax) | Up to 3 Years
  Phase 1a/1b - Sampling following the first dose, pre and post-dose at selected cycles, and at the end of treatment
PK parameters of NX-1607: volume of distribution | Up to 3 Years
  Phase 1a/1b - Sampling following the first dose, pre and post-dose at selected cycles, and at the end of treatment
PK parameters of NX-1607: half-life and time to maximum plasma concentration | Up to 3 Years
  Phase 1a/1b - Sampling following the first dose, pre and post-dose at selected cycles, and at the end of treatment
PK parameters of NX-1607: accumulation ratio (Racc) | Up to 3 Years
  Phase 1a/1b - Sampling following the first dose, pre and post-dose at selected cycles, and at the end of treatment
PD Biomarkers: Changes from baseline in inflammatory cytokine expression in the circulating immune cells | Up to 3 Years
  Phase 1a/1b - Sampling following the first dose, pre and post-dose at selected cycles, and at the end of treatment
Objective response rate (ORR) per disease-specific response criteria as assessed by the Investigator | Up to 3 Years
  Phase 1a
Duration of response (DOR) as assessed by the Investigator | Up to 3 Years
  Phase 1a/1b
Disease control rate (DCR) as assessed by the Investigator | Up to 3 Years
  Phase 1a/1b
Progression-free survival (PFS) as assessed by the Investigator | Up to 3 Years
  Phase 1a/1b
Overall survival (OS) as assessed by the Investigator | Up to 3 Years
  Phase 1a/1b
Incidence of TEAEs, including Grade ≥ 3 TEAEs, treatment emergent SAEs, TEAEs leading to study drug discontinuation, and deaths due to TEAEs | Up to 3 Years
  Phase 1b
Time to disease progression assessed by the Investigator (according to relevant disease histology) | Up to 3 Years
  Phase 1b
Incidence of IrAEs and all deaths | Up to 3 Years
  Phase 1b
Time from start of treatment to disease progression based on PCWG3 criteria | Up to 3 Years
  Phase 1b (mCRPC cohort only)
PD Biomarkers: Changes from baseline in tumor tissue biopsies of immune cell infiltration or other histological features | Up to 3 Years
  Phase 1b

CONTACTS AND LOCATIONS:
Overall Officials: Linda Neuman, MD, Study Director — Nurix Therapeutics, Inc.
Locations (17):
- United States (10):
  - City of Hope, Duarte, California
  - University of Southern California, Los Angeles, California
  - University of California, San Francisco, San Francisco, California
  - University of Colorado School of Medicine, Aurora, Colorado
  - University of Chicago, Chicago, Illinois
  - University of North Carolina, Chapel Hill, North Carolina
  - University of Oklahoma, Oklahoma City, Oklahoma
  - MD Anderson Cancer Center, Houston, Texas
  - University of Virginia, Charlottesville, Virginia
  - Fred Hutchinson Cancer Center, Seattle, Washington
- United Kingdom (7):
  - Royal Marsden Hospital NHS Foundation Trust, Sutton, Surrey
  - Addenbrookes Cambridge University Hospital, Cambridge
  - Beatson West of Scotland Cancer Centre, Glasgow
  - Sarah Cannon Research Institute, London
  - The Christie NHS Foundation Trust, Manchester
  - Northern Centre for Cancer Care, Newcastle
  - Churchill Hospital, Oxford

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wolf D, Baier G. IFNgamma Helps CBLB-Deficient CD8+ T Cells to Put Up Resistance to Tregs. Cancer Immunol Res. 2022 Apr 1;10(4):370. doi: 10.1158/2326-6066.CIR-22-0080. PMID 35362047